CLINICAL TRIAL: NCT06413368
Title: Maralixibat in Patients With Cystic Fibrosis and Constipation, A Within-Subjects Pilot Study
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Jaya Punati, Medical Staff/USC Faculty CWR, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-23-00352
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Constipation Chronic Idiopathic; Cystic Fibrosis
Keywords: Maralixibiat; Cystic Fibrosis; Chronic Constipation; Bristol Stool
MeSH Terms: conditions — Cystic Fibrosis | interventions — maralixibat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment arm (Other): within - subjects study
  Interventions: Drug: Maralixibat 9.5 MG/ML [Livmarli]

INTERVENTIONS:
Drug: Maralixibat 9.5 MG/ML [Livmarli] — Within Study subjects receiving 2 weeks of treatment with Maralixibat 9.5 MG/ML [Livmarli] and compare to baseline treatment.

SUMMARY:
Chronic constipation is a feature of children with cystic fibrosis (CF). This is postulated to be a result of inhibition of secretory activity of the gastrointestinal luminal cells due to ineffective chloride channel function. Typical laxatives that work as osmotic agents fail to produce adequate relief in this population.

Maralixibat is a non-systemic bile acid transport inhibitor (IBATi) that acts by interrupting bile acid reabsorption in the ileum thus interrupting the normal enterohepatic circulation. This interruption results in a larger volume of bile acids reaching the colon and being excreted in stool. Bile acids are known to decrease bowel transit time, increase mucosal permeability and secretions, as well as alter gut microbiota resulting in diarrhea.

The overarching hypothesis of the study is that Maralixibat will improve stool consistency in children (Age <18 years) with cystic fibrosis and constipation (Bristol Stool Scale <4). Specifically, we aim to test the hypothesis that IBATi improves the consistency of stool to Bristol scale >4 in children with CF and constipation.

We will recruit a total of 20 patients with CF and constipation (defined as Bristol Stool Scale <4 for 1 week prior to enrollment while on a stable laxative regimen for at least 4 weeks.) Design is a 'Within-Subjects' study by which each enrolled patient will take Maralixibat for 2 weeks total in addition to their stable laxative regimen during the study. Stool consistency & ease of defecation will be recorded before and during the study period by families of enrolled patients via materials provided by the investigators. Stool consistency and ease of defecation will be compared before and after initiation of Maralixibat.

The primary endpoint: Improvement in stool consistency to Bristol scale >4 in children with CF and constipation. The secondary endpoint: Improvement in ease of defecation in children with CF and constipation. This will be measured via survey using a standardized scale (Bristol Stool Scale) and questionnaires developed by the research team. Analysis will involve comparison of pre-intervention to post-intervention stool consistency & survey

DETAILED DESCRIPTION:
Study Title Maralixibat in Patients with Cystic Fibrosis and Constipation, A Within-Subjects Pilot Study Objectives Primary Objective: The primary aim of the study is to assess improvement in stool consistency in children (1 - 18 years of age) with cystic fibrosis. We will recruit a total of 20 patients with CF and constipation. Constipation will be defined as Bristol Stool Scale of < 3 for 1 week prior to enrollment while on a stable laxative regimen for at least 4 weeks. They will receive Maralixibat for 3 weeks. Questionnaires via REDCap survey will be administered by the investigators pre- and post-intervention to assess changes in stool consistency and frequency after adding Maralixibat to their constipation regimen.

Secondary Objective: The secondary aims include assessment for improved ease of defecation (as subjectively judged by patients & their parents) after adding Maralixibat to their constipation regimen. Questionnaires via REDCap survey will be administered by the investigators pre and post intervention to assess changes in ease of defecation after adding Maralixibat to their constipation regimen.

Design and Outcomes This study is a Within-Subjects Clinical Pilot study to examine the effect Maralixibat has on constipation in children (1 - 18 years of age) with cystic fibrosis (CF). We will recruit a total of 20 patients with CF and chronic constipation (defined as Bristol stool scale of < 3 for 1 week prior to enrollment while on stable medication regimen for at least 4 weeks). They will receive IBATi for 3 weeks in addition to their stable conventional constipation medication regimen. Questionnaires via REDCap survey will be administered by the investigators pre and post intervention to assess changes in stool consistency, frequency, and ease of defecation after adding Maralixibat to their constipation regimen.

Estimated Study Timelines:

* The duration of an individual subject's participation in the study: 3 weeks
* The duration anticipated to enroll all study subjects: 2 years
* The estimated date for the investigators to complete this study (complete primary analyses): 30 months Interventions and Duration This study will compare a conventional constipation regimen for chronic constipation (stool softeners, stimulant laxatives, dietary changes, etc.) to conventional constipation regimen + Maralixibat.
* Conventional Constipation Regimen: Stable regimen for at least 4 weeks
* Conventional Constipation Regimen + Maralixibat: 3 weeks

Sample Size and Population Target Population: Children (1 - 18 years of age) with Cystic Fibrosis & Chronic Constipation (defined as Bristol stool scale of < 3 for 1 week prior to enrollment while on stable medication regimen for at least 4 weeks).

Number of Participants: 20

This is a Within-Subjects study design, so there will not be randomization and all patients will receive the study intervention. The period prior to initiation of Maralixbat with serve as the 'baseline' or 'control' of our primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1-18 years Proven diagnosis of Cystic Fibrosis (via genetic testing or sweat chloride testing) Proven diagnosis of Chronic constipation (Bristol stool scale rating of < 3 while on stable conventional therapy regimen) On stable (no medication changes or dose adjustments) conventional constipation medication regimen for chronic constipation (stool softeners, stimulant laxatives, dietary interventions) for at least 4 weeks.

Exclusion Criteria:

* The following are exclusion criteria for our study. All candidates meeting any of the exclusion criteria at baseline will be excluded from study participation:

Uncontrolled fat-soluble vitamin deficiency (Vitamin A, E, D, or K) Changes to conventional constipation medication regimen <4 weeks prior to initiation of Maralixibat Adequately treated chronic constipation on conventional regimen (Bristol stool scale rating of > 3) Allergy or sensitivity to the study drugs or their ingredients Inability or unwillingness of individual or legal guardian/representative to given written informed consent.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in stool consistency by 1 point in Bristol scale or transition to Bristol scale > 3 after study drug | baseline to 3 weeks
  Constipation is defined as stool consistency of Bristol Scale 1 to 3. Our primary endpoint is looking for a change of 1 unit of the scale or transition to a scale of >3

SECONDARY OUTCOMES:
Change in subjective scoring in ease of stooling with the addition of Maralixibat to a conventional constipation medication regimen via subjective questionnaire. | Baseline - 3 weeks
  Maralixibat inhibits baseline absorption which in turn results in looser stools by osmosis.
  We will use a questionnaire to record subjective report of ease of stooling by patients from baseline prior to intervention using a Likert score of 1-5
  1. - cannot stool
  2. - Difficulty stooling
  3. - neither easy nor difficult
  4. - Easier stooling with medication
  5. - No issues with stooling

CONTACTS AND LOCATIONS:
Overall Officials: Jaya Punati, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No